CLINICAL TRIAL: NCT00883194
Title: A Single-center, Randomized, Placebo-controlled, Double-blind, Single-dose, Efficacy of PRF-108 4% and PRF-110 4% Versus Ropivacaine Solution 0.5% in an Experimental Pain Model
Brief Title: A Safety and Effectiveness Pilot Study of PRF-108 and PRF-110 in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PainReform LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRF108-POC99-09
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Pain
Keywords: Experimental Pain Model
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): PRF-108 Gel, 4% ropivacaine
  Interventions: Drug: PRF-108
- 2 (Placebo Comparator): PRF-108 Gel, Vehicle
  Interventions: Drug: Placebo
- 3 (Active Comparator): Ropivacaine Solution 0.5%
  Interventions: Drug: Ropivacaine
- PRF-110, 4% (Experimental): PRF-110, 4% ropivacaine
  Interventions: Drug: PRF-110

INTERVENTIONS:
Drug: PRF-108 — Ropivacaine
  Arms: 1
Drug: Placebo — PRF-108 Placebo
  Arms: 2
Drug: Ropivacaine — Solution
  Arms: 3
Drug: PRF-110
  Other Names: ropivacaine
  Arms: PRF-110, 4%

SUMMARY:
This is a clinical study testing PRF-108 and PRF-110 (a new extended release 4% gel formulations of ropivacaine) in an experimentally induced pain model in healthy volunteers. PRF-108 and PRF-110 are designed to deliver slow release of ropivacaine over 72 hours.

DETAILED DESCRIPTION:
This is a clinical study testing PRF-108 and PRF-110 (a new extended release 4% gel formulations of ropivacaine) in an experimentally induced pain model in healthy volunteers. PRF-108 and PRF-110 are designed to deliver slow release of ropivacaine over 72 hours.

The purpose of this study is to investigate the safety (side effects if any occurs) associated with the single administration of PRF-108 or PRF-110 and evaluate their analgesic effect in an experimentally induced pain model compared with ropivacaine Solution 0.5% and Vehicle Gel.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects between 18-60 years of age;
2. Subjects are within ±10% of ideal body weight/height (based on frame size) as given by the Metropolitan Life Insurance Tables;
3. Subjects are ASA Category I and in normal physical health as judged by physical and laboratory examinations and have a negative urine based screen for drugs of abuse;
4. Subjects must agree to refrain from ingesting any analgesic medication for 3 days or 5 half-lives of the drug prior to and during the study period and alcohol for 1 day prior to and during the study period;
5. Subjects can tolerate a 0.5mL injection of saline in the lower back area.
6. The subject is capable of reading, comprehending, and signing the informed consent form.

Exclusion Criteria:

1. Subjects with a history of any significant hepatic, renal, endocrine, cardiac, neurological, psychiatric, gastrointestinal, pulmonary, hematologic, or metabolic disorders, including glaucoma, diabetes, emphysema, and chronic bronchitis;
2. Subjects with a history of any type of cancer;
3. Subjects with conditions that affect the absorption, metabolism, or passage of drugs out of the body, (e.g., sprue, celiac disease, Crohn's disease, colitis, or liver, kidney, or thyroid conditions);
4. Subjects with any history of alcohol or substance abuse (including a positive drug screen test);
5. Subjects that currently have or have a history of hypertension;
6. Subjects with a known hypersensitivity to any local anesthetic drug;
7. Subjects with a history of benign prostatic hyperplasia or difficulty in urination;
8. Subjects with a hematocrit level below the normal range on the screening laboratory examination;
9. Subjects with any clinically significant abnormal lab result (as judged by the Principal Investigator);
10. An abnormal ECG at screening including PR>200 ms, QRS>110 ms, QTcF<380 or >400 ms, lead II T wave abnormalities. Non-specific T wave abnormalities in leads other than lead II are permissible if not accompanied by any other morphological abnormalities.
11. Subjects with any condition or history felt by the Investigator to place the subject at increased risk;
12. Subjects who have smoked or chewed tobacco-containing substances within 6 months prior to the start of the study;
13. Subjects judged by the Investigator to be unable or unwilling to comply with the requirements of the protocol;
14. Subjects who have used an investigational drug within 30 days prior to entering the study;
15. Subjects who have donated blood within 3 months prior to the start of the study (including blood donation related to the surgical procedure);
16. Subjects who have previously participated in the trial;
17. Subjects who are members of the study site staff directly involved with the study or a relative of the Sponsor or other personnel involved with the study.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The duration of analgesia | 3 days

SECONDARY OUTCOMES:
PRF-108 and PRF-110 Safety | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Naveh, Study Chair — PainReform LTD
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel